CLINICAL TRIAL: NCT02676310
Title: Dose Escalation Study of the Safety, Tolerability, and Pharmacokinetics of Bimatoprost Topical Solution in the Treatment of Androgenetic Alopecia in Men
Brief Title: Safety, Tolerability, and Pharmacokinetics of Bimatoprost in Men With Androgenetic Alopecia (AGA)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 192024-085
Record Dates: First submitted 2016-02-04; First posted 2016-02-08 (Estimated); Last update posted 2017-03-17 (Actual); Status verified 2017-03

CONDITIONS: Alopecia; Alopecia, Androgenetic; Baldness
MeSH Terms: conditions — Alopecia | interventions — Bimatoprost

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Cohort 1: Bimatoprost 0.3% (Formulation B) (Experimental): 0.25 mL of bimatoprost 0.3% (Formulation B) applied onto pre-specified area on the scalp once daily for 28 days.
  Interventions: Drug: Bimatoprost
- Cohort 2: Bimatoprost 1% (Formulation A) (Experimental): 0.25 mL of bimatoprost 1% (Formulation A) applied onto pre-specified area on the scalp once daily for 28 days.
  Interventions: Drug: Bimatoprost
- Cohort 2: Bimatoprost 1% (Formulation B) (Experimental): 0.25 mL of bimatoprost 1% (Formulation B) applied onto pre-specified area on the scalp once daily for 28 days.
  Interventions: Drug: Bimatoprost
- Cohort 3: Bimatoprost 1% (Formulation B) (Experimental): 1 mL of bimatoprost 1% (Formulation B) applied onto pre-specified area on the scalp once daily for 28 days.
  Interventions: Drug: Bimatoprost
- Cohort 4: Bimatoprost 3% (Formulation B) (Experimental): 1 mL of bimatoprost 3% (Formulation B) applied onto pre-specified area on the scalp once daily for 28 days.
  Interventions: Drug: Bimatoprost

INTERVENTIONS:
Drug: Bimatoprost
  Other Names: Bimatoprost Solution applied onto pre-specified area on the scalp daily for 28 days.

SUMMARY:
This is a safety, tolerability, and pharmacokinetics study of bimatoprost in male patients with androgenetic alopecia (AGA).

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate male pattern baldness (androgenic alopecia) with ongoing hair loss for at least 1 year

Exclusion Criteria:

* History of Paget's disease, osteoporosis, or bone malignancy
* History of bone fracture within the previous 12 months, except for metatarsal, metacarpal, or skull fractures
* Patient is currently undergoing radiation therapy or anticipates undergoing radiation therapy at any time during the study
* Drug or alcohol abuse within 12 months
* HIV positive
* Received hair transplants or had scalp reductions
* Use of hair weaves, hair extensions or wigs within 3 months
* Application of topical medications, minoxidil or nonsteroidal anti-inflammatory drugs (NSAIDs) to scalp within 4 weeks

Ages: 18 Years to 49 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2016-03; Primary Completion 2017-01 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Treatment Emergent Adverse Events (TEAEs) | 42 Days
Change from Baseline in Local Dermal Tolerability as Assessed by the Subject Using a 4-Point Scale | Baseline, 42 Days
Maximum plasma level (Cmax) of bimatoprost and its acid metabolite | 31 Days

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (3):
- United States (3):
  - DermResearch, LLC, Austin, Texas
  - J&S Studies Inc., College Station, Texas
  - E&R Research Foundation, Lynchburg, Virginia